CLINICAL TRIAL: NCT00536627
Title: Randomised, Opened, Multicentre Phase I/II Trial in Patients With Chronic Hepatitis B With HBV VL < 12 IU/ml and Under Treatment With NRTI, Which Evaluated Efficacy and Tolerance of Vaccination With Naked DNA on Viral Replication After Analogs' Treatment Interruption. ANRS HB02 VAC-ADN
Brief Title: Efficacy and Tolerance of Naked DNA Vaccine in Patients With Chronic B Hepatitis
Acronym: VAC-ADN
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: French National Agency for Research on AIDS and Viral Hepatitis (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2007-001682-15; ANRS HB02 VAC-ADN
Record Dates: First submitted 2007-09-26; First posted 2007-09-28 (Estimated); Last update posted 2011-12-19 (Estimated); Status verified 2011-12

CONDITIONS: Chronic Hepatitis B
Keywords: DNA vaccine
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Patients will receive 5 injections of DNA vaccine at weeks 0, 8, 16, 40, 44.
  Interventions: Biological: DNA vaccine pCMVS2.S
- 2 (No Intervention)

INTERVENTIONS:
Biological: DNA vaccine pCMVS2.S — Patients will receive injections of 1 ml of vaccine (1 mg/ml) at weeks 0, 8, 16, 40 and 44
  Arms: 1

SUMMARY:
The purpose of this study is to determine if DNA vaccination of chronic HBV patients under treatment with NRTI can restore T-cell responsiveness and delay virologic reactivation after treatment discontinuation.

DETAILED DESCRIPTION:
Despite the availability of effective vaccines against hepatitis B, over 370 million people worldwide remain persistently infected with HBV. Persistent infection is associated with chronic liver disease that can lead to the developement of cirrhosis and hepatocellular carcinoma in two-third of persons. Treatment of chronic hepatitis B relies on the use of analogs such as lamivudine, adefovir, entecavir or immunostimulators such as interferons. Although analogs are efficient, genotypic resistance occurs after one year of treatment and the rate of virologic relapse is high after treatment discontinuation.

HBV is a non cytopathic virus and liver damage is caused by immune response against infected hepatocytes and to a non specific inflammatory response. Immune response contributes to the virus clearance. In acute hepatitis B infection, T cell response is polyclonal, specific and vigorous, whereas in patients with chronic infection, responses remain weak, less specific and hardly detectable in peripheral blood.

T cell responses could be induced or restored by antigenic stimulation such as vaccination. In a previous phase I clinical trial, we showed that DNA vaccination with plasmid pCMVS2.S is safe and can specifically, but transiently activate T-cell responses in chronic HBV-carriers not responding to current antiviral therapies.

Analogs such as lamivudine and adefovir were shown to enhance T cell responses concomitantly with viral load decrease. In this phase I/II clinical trial, we would like to determine if DNA vaccination of chronic HBV patients under treatment with NRTI can restore T-cell responsiveness and delay virologic reactivation after treatment discontinuation.

ELIGIBILITY:
Inclusion Criteria:

* chronic hepatitis B with or without AgHBe
* no cirrhosis and no hepatocellular carcinoma
* treatment with NRTI unchanged for at least 3 months
* undetectable HBV viral load for 12 months
* HBV viral load < 12 IU/ml at screening
* sGPT < 5N
* tetanus immunization or booster dose for less than 8 years
* accurate birth control or menopausal women or sterility
* sickness insurance
* signed informed consent

Exclusion Criteria:

* HLA-DR 15/16
* coinfections with HDV, HCV and/or HIV
* treatment with immunomodulators
* immunosuppressors
* long-term corticotherapy (over 4 weeks)
* active intravenous drug-users
* prolonged and excessive consumption of alcohol (men > 40g/day ; women > 30g/day ; for more than 5 years)
* medical history of autoimmune disease or presence of autoantibodies
* previous immunization by HBV vaccine of less than 5 years
* previous immunization by DNA vaccine against HBV
* personal or family medical history of demyelinising diseases
* uncontrolled hypophosphatemia
* renal failure, renal transplantation, haemodialysis
* pregnancy, breast-feeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2008-01; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Primary endpoint is virologic failure defined by 1) reactivation after analogs' treatment interruption, 2) virologic breakthrough during treatment with analogs, 3) the impossibility for the patients to interrupt treatment at week 48 | at week 72

SECONDARY OUTCOMES:
Delay of appearance of virologic failure | at Week 72
Biological and clinical tolerance of DNA vaccine | all along the trial
Immunological responses | At weeks 18, 40, 46, 60, 72
Clinical progression of hepatitis B | all along the trial

CONTACTS AND LOCATIONS:
Overall Officials: Hélène FONTAINE, MD, Principal Investigator — Pôle d'Hépatologie, Hôpital COCHIN, PARIS, FRANCE; Jean-Pierre ABOULKER, MD, Study Chair — INSERM SC-10, VILLEJUIF, FRANCE
Locations (1):
- FONTAINE Hélène, Paris, France

REFERENCES:
- [Background] Mancini-Bourgine M, Fontaine H, Brechot C, Pol S, Michel ML. Immunogenicity of a hepatitis B DNA vaccine administered to chronic HBV carriers. Vaccine. 2006 May 22;24(21):4482-9. doi: 10.1016/j.vaccine.2005.08.013. Epub 2005 Aug 18. PMID 16310901
- [Background] Mancini-Bourgine M, Fontaine H, Scott-Algara D, Pol S, Brechot C, Michel ML. Induction or expansion of T-cell responses by a hepatitis B DNA vaccine administered to chronic HBV carriers. Hepatology. 2004 Oct;40(4):874-82. doi: 10.1002/hep.20408. PMID 15382173
- [Derived] Fontaine H, Kahi S, Chazallon C, Bourgine M, Varaut A, Buffet C, Godon O, Meritet JF, Saidi Y, Michel ML, Scott-Algara D, Aboulker JP, Pol S; ANRS HB02 study group. Anti-HBV DNA vaccination does not prevent relapse after discontinuation of analogues in the treatment of chronic hepatitis B: a randomised trial--ANRS HB02 VAC-ADN. Gut. 2015 Jan;64(1):139-47. doi: 10.1136/gutjnl-2013-305707. Epub 2014 Feb 20. PMID 24555998
- [Derived] Godon O, Fontaine H, Kahi S, Meritet JF, Scott-Algara D, Pol S, Michel ML, Bourgine M; ANRS HB02 study group. Immunological and antiviral responses after therapeutic DNA immunization in chronic hepatitis B patients efficiently treated by analogues. Mol Ther. 2014 Mar;22(3):675-684. doi: 10.1038/mt.2013.274. Epub 2013 Dec 5. PMID 24394187